CLINICAL TRIAL: NCT05254938
Title: The Halland Obesity Municipal Effort for Children
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Region Halland (Other)
Responsible Party: Sponsor
Other Study IDs: 4294300
Record Dates: First submitted 2021-10-22; First posted 2022-02-24 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Childhood Obesity; Physical Inactivity; Physical Activity; BMI; Neurodevelopmental Disorders; Hypertension
MeSH Terms: conditions — Pediatric Obesity; Sedentary Behavior; Motor Activity; Neurodevelopmental Disorders; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: The Halland Obesity Municipal Effort for children — A comprehensive, intensive lifestyle intervention for the children with the greatest need of intensive treatment.

SUMMARY:
A retrospective study to investigate the method called The Halland Obesity Municipal Effort for children. All children participating in the intervention since the start of this specific method will be eligible for inclusion. The aims are to describe participants and the method-specific activities they are participating in, as well as the effect on their health and school grades.

DETAILED DESCRIPTION:
This method involves the entire municipal community in Laholm and Kungsbacka (two cities in Sweden): Pediatric care unit, Child Psychiatry, Social services, School healthcare, private companies, and local sports clubs. The model includes group activities and individual activities and offer 15 different health promoting and free activities per week.

All activities are modified and take place in a safe environment. The activities range from golf, riding, gym training, swimming, fishing, art classes, karate, dance classes, and the possibility for the child to get a grade in Physical Education through a specific collaboration with the local schools in the municipality.

The children are given a fruit at each activity and cooking classes are frequently given. The municipal activity coordinator who is responsible uses different methods such as KASAM, Health Action Model and Empowerment to help each child develop skills in self-monitoring, goal setting, problem solving, contingent reward systems, and stimulus control. Parents are given a specific support program called COPE, Community Parent Education. Some activities include the whole family.

In addition to the weekly activities, the activities are also always given on school holidays and weekends when children are known to be less active.

This study will investigate this method by focusing on BMI, metabolic control, blood pressure, level of physical activity, age, sex, the existence of comorbidities, presence of neurodevelopmental disorders, school related issues, involvement of social services, need of grades in Physical Education and help to learn how to swim, which activities the children were undertaking as well as the frequency of participation. The proportion of children achieving full 12 years of education will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients involved in the HOME project since the start. Children that have been offered this intense intervention.

Exclusion Criteria: Those who are not willing to participate.

-

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — We will follow the gender that the patient aknowledges based on regional ethical considerations.
Study Population: Children aged 5-21 that were followed at a pediatric clinic for obesity and with complicating factors such as comorbidity, socioeconomic vulnerability, lonliness and problematic school absenteeism.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
12 years completed education | At the age of 19.
  Registry data regarding completion of 12 school years, will be assessed for each patients at the age of 19.
Change from baseline in BMI after 6 month | Baseline and month 6.
  BMI (weight/height^2), obtained from health records at interventions start and after 6 months of intervention.
Change from baseline in BMI after 12 month | Baseline and month 12.
  BMI (weight/height^2), obtained from health records at interventions start and after one year of intervention.
Change from baseline in BMI after 18 months | Baseline and month 18.
  BMI (weight/height^2), obtained from health records at interventions start and after 18 months of intervention.
Change from baseline in gucose homeostasis | Baseline and month 12.
  Blood samples concerning blood sugar levels (HbA1c, fasting glucose, insulin). Obtained from health records at interventions start and after one year of intervention.
Change from baseline in blood pressure | Baseline and month 12.
  Blood pressure (mm/Hg) measured in right arm sitting down after 5 minutes of rest. Obtained from health records at interventions start and after one year of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Josefine Roswall, MD, PhD, Study Chair — Region Halland
Locations (1):
- Lovisa Sjögren, Särö, Sweden